CLINICAL TRIAL: NCT07141771
Title: An Umbrella Study of Recurrent, Extensive Stage Small Cell Lung Cancer Based on Molecular Typing
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UM-SCLC
Record Dates: First submitted 2025-07-31; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: SCLC, Extensive Stage
MeSH Terms: interventions — fluzoparib; Topotecan; Etoposide; PM 01183; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- N subtype (Experimental): N subtype
  Interventions: Drug: Serplulimab; Drug: Topotecan/Irinotecan/Paclitaxel/Temozolomide
- subtype P and subtype A with low BCL-2 expression (Experimental): subtype P and subtype A with low BCL-2 expression
  Interventions: Drug: Fluzoparib; Drug: Temozolomide
- subtype Y (Experimental): subtype Y
  Interventions: Drug: Serplulimab; Drug: Topotecan/Irinotecan/Paclitaxel/Temozolomide
- low expression in SLFN11 (Experimental): low expression in SLFN11
  Interventions: Drug: Serplulimab; Drug: Etoposide/Carboplatin/Cisplatin
- high expression in SLFN11 (Experimental): high expression in SLFN11
  Interventions: Drug: Serplulimab; Drug: Lurbinectedin

INTERVENTIONS:
Drug: Serplulimab — Serplulimab: 4.5mg/kg, ivgtt, 21 days/cycle
  Other Names: HLX10; Hetronifly
  Arms: N subtype; high expression in SLFN11; low expression in SLFN11; subtype Y
Drug: Fluzoparib — 100mg BID oral
  Other Names: HS-10160; HR011417; SHR3162; SHR133162
  Arms: subtype P and subtype A with low BCL-2 expression
Drug: Topotecan/Irinotecan/Paclitaxel/Temozolomide — second-line chemotherapy options: Topotecan/Irinotecan/Paclitaxel/Temozolomide etc.
  Arms: N subtype; subtype Y
Drug: Etoposide/Carboplatin/Cisplatin — First-line chemotherapy: the original first-line chemotherapy regimen, recommended Etoposide 100mg / m2 d1-3, Carboplatin AUC = 5 d1 / Cisplatin 75mg / m2 d1 q21d
  Arms: low expression in SLFN11
Drug: Lurbinectedin — 2.6mg/m2 (3 patients, if safe, in the 3.2mg / m2 dose group) or 3.2 mg / m2, ivgttd,21d / cycle .
  Other Names: PM01183; Zepzelca
  Arms: high expression in SLFN11
Drug: Temozolomide — 150mg/m2, oral, on days 1-5,28d / cycle
  Arms: subtype P and subtype A with low BCL-2 expression

SUMMARY:
Small-cell lung cancer (SCLC) has a high degree of malignancy and extremely poor prognosis, slow progress in the treatment of ES-SCLC, and a more ideal posterior therapy needs to be explored. This is an I / II, phase umbrella study to explore afterline treatment options following progression of frontline platinum-containing therapy for small cell lung cancer.

This study includes 2 parts:

Part 1 will enroll patients with end of first-line platinum-containing therapy and progression interval of less than 180 days or more of second-line therapy (no first-line relapse time required).

Part 2 will enroll patients with end of first-line platinum-containing therapy greater than 180 days.

Based on the optimal selection of patients with recurrent broad-stage small cell lung cancer with different molecular and clinical characteristics, we further explored different treatment modes suitable for different populations through umbrella cohort studies.

DETAILED DESCRIPTION:
Small-cell lung cancer (SCLC) has a high degree of malignancy and extremely poor prognosis, slow progress in the treatment of ES-SCLC, and a more ideal posterior therapy needs to be explored. This is an I / II, phase umbrella study to explore afterline treatment options following progression of frontline platinum-containing therapy for small cell lung cancer.

This study includes 2 parts:

Part 1 will enroll patients with end of first-line platinum-containing therapy and progression interval of less than 180 days or more of second-line therapy (no first-line relapse time required).

Cohort 1 patients enrolled with N subtype were given either Serplulimab plus second-line chemotherapy or other treatment as assessed by the physician; cohort 2 patients enrolled with subtype P and subtype A with low BCL-2 expression were given Fluzoparib with Temozolomide ; cohort 3 patients enrolled with subtype Y received Serplulimab plus second-line chemotherapy ;

Part 2 will enroll patients with end of first-line platinum-containing therapy greater than 180 days.

Cohort 4 patients with low expression in SLFN11 were given Serplulimab plus first-line chemotherapy ; cohort 5 patients with high SLFN11 expression were given Serplulimab plus Lurbinectedin.

Based on the optimal selection of patients with recurrent broad-stage small cell lung cancer with different molecular and clinical characteristics, we further explored different treatment modes suitable for different populations through umbrella cohort studies, which is of great significance to prolong the survival of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to fully understand and sign the informed consent form, including compliance with the requirements and restrictions listed in the ICF and this protocol. A legally authorized representative may sign off on behalf of the subject.

2. Subject age must be 18 years (including 18 years). 3. Participants must have stage IV metastatic small cell lung cancer confirmed by histology or cytology, not suitable for radical surgery or radiotherapy, and have disease progression after first-line standard platinum-containing regimen.

4. The ECOG / WHO fitness status score is 0 to 1. 5. Expected survival time must be at least 12 weeks. 6. Participants agreed to perform the biopsy and could obtain enough tissue specimens for whole-exon sequencing, transcriptome sequencing, and multiplex fluorescent immunohistochemical detection.

7.The patient has sufficient important organ functions during screening (requiring no blood transfusion, no use of hematopoietic stimulating factors or human albumin preparations within 14 days prior to screening), and the specific definition is as follows:

1. Blood routine: Absolute neutrophil count (Absolute neutrophil count, ANC) 1.5109 / L; Platelet Count (Platelet, PLT)≥100×109/L; Hemoglobin content (Hemoglobin, HGB) 90 g / L;
2. liver function: serum total bilirubin (Total bilirubin, TBIL) 1.5 Upper Normal Value (Upper limit of normal value, ULN), Patients with liver metastasis or with proven Gilbert syndrome, TBIL≤3×ULN. For subjects without liver metastases, Alanine aminotransferase (Alanine aminotransferase, ALT) and aspartate aminotransferase (Aspartate transferase, AST) ≤2.5×ULN, Subjects with liver metastases, ALT or AST 5 ULN;
3. Renal function: creatinine clearance calculated according to the Cockcroft-Gault method (Clearance of creatinine, CCr) 60 mL/min;
4. Coagulation: activated partial thromboplastin time (Activated partial thromboplastin time, APTT) and the international standardized ratio (International normalized ratio, INR) 1.5 ULN (subjects receiving anticoagulation are within treatment range);
5. cardiac function criteria: echocardiogram (Echocardiography, ECHO) showed a left ventricular ejection fraction (LVEF) greater than 50%.

   8. The blood pregnancy test must be negative within 7 days before the first use of the test drug; fertile qualified patients (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) with their partner during the trial and at least 6 months after the last dose. Ferproductive patients were defined as sexually mature and with biologically underlying fertility.

   9. Crias for molecular typing selection:
   1. characteristics of transcription factor subtypes:
   2. (1) SCLC-A and N types belong to neuroendocrine types, and SCLC-P and-I are cells with non-neuroendocrine subtypes. SCLC-A and N had significantly higher expression of neuroendocrine markers (chromaffin A (CgA) and synaptic vesicle protein (Syn)), while SCLC-P and I highly expressed the neuroendocrine inhibitory gene RE1 silent transcription factor (REST).
   3. (2) SCLC-I is the most characteristic of stromal cells, while SCLC-A has the most characteristic of epithelial cells. High expression markers of SCLC-I of stromal cells: VIM and AXL. Most of the SCLC cells expressing the thyroid transcription factor (TTF 1) belong to the SCLC-A type.
   4. (3) The vast majority of TP 53 and RB 1 mutations do not differ in subtype classification, and the classification of subtypes is not associated with specific gene mutations.
   5. In conclusion, SCLC-A is neuroendocrine with epithelial cells, expressing TTF 1; SCLC-N, also neuroendocrine, but not TTF 1; SCLC-P and SCLC-I are non-neuroendocrine, while SCLC-I has a subtype characterized by mesenchymal cells.
   6. H-score method (integral system): IHC test of tissue specimens to calculate the product of the percentage of positive tumor cell nuclear staining (0-100%) observed under the optical microscope and its staining intensity (intensity, 0,1 +, 2 +, 3 +), to obtain H-score (range 0-300) 13.
   7. SLFN11:1 + under IHC score is positive 13, and the cut-off value is usually selected 10,10, which is defined as high expression 28.
   8. BCL-2: The average copy number per spot was calculated based on the minimum and maximum number of Bcl-2 FISH signal from each nucleus in each tissue site. Copy arrays were constructed based on the absolute gene copy number using the following criteria: 1 to 2 signals with average copy number <2.5; 3 to 4 signals, average copy number 2.5 and <4.5; 5 to 6 signals, average copy number 4.5 and <6.5; and 7 to 10 signals, with average copy number 6.5 29.
   9. c-Myc: IHC 1 +, 2 + and 3 + were positive; 0 was negative.
   10. If two or more markers in the same class have an H score of more than 10, then multiple markers in the tumor may be positive. The predominant marker was defined as the marker with the highest H-Score.
   11. TROP-2: IHC stains at least 10% of tumor cells with an intensity score of 1 + (weak), and 2 + (moderate) and 3 + (strong) are defined as positive 22. At the same time, ANPY will be tested simultaneously (before the start of treatment) and submitted for transcriptomic testing.

   10, with at least 1 measurable lesion according to RECIST 1.1.

   Exclusion Criteria:
   1. Acute toxicity associated with prior anti-tumor therapy for 4 weeks prior to the first dose did not return to grade NCI CTCAE v5.0 1 or the baseline level specified by the entry criteria (excluding alopecia or fatigue).
   2. The following drugs or herbal supplements cannot be stopped within 3 weeks before and during the study: (1) strong inducers or inhibitors of CYP3A4; (2) drugs mainly metabolized by CYP3A4;
   3. The subject does not agree to secondary biopsy or cannot obtain enough tissue specimens for full exon sequencing, transcriptome sequencing, and multiple fluorescent immunohistochemical testing.
   4. Mean corrected QT interval (Corrected QT interval, QTc, Fridericia's correction) from 12-lead ECG (12-Electrocardiograph, ECG)> 470 ms (3 repeats). Various clinically significant cardiac rhythm, conduction, and resting ECG morphology abnormalities, such as complete left bundle branch block, degree III conduction block, degree II conduction block, and PR interval> 250 ms. Various factors that may increase the risk of QTc extension or arrhythmic events, such as cardiac failure, hypokalemia, congenital long QT syndrome, long QT syndrome in immediate family history or unexplained sudden death under 40 years of age, are using any medication with known QT interval extension.
   5. Acute or chronic active hepatitis B [defined as hepatitis B surface antigen (HbsAg) and/or hepatitis B core antibody (HbcAb) positive and hepatitis B virus (HBV) DNA copy number ≥ 1 × 10]3 copies per mL or ≥ 200 IU/mL.
   6. Acute or chronic active hepatitis C (HCV), or HCV antibody positive and HCV-RNA levels greater than the upper central reference limit.

   7 Patients with active brain metastases are enrolled if their central nervous system (Central nervous system, CNS) tumor metastasis is limited to supratentorial or cerebellum, is adequately treated (surgery or radiotherapy), has maintained radiographic stability for at least 4 weeks, and does not require corticosteroids to control symptoms.

   8 Concurrent diseases failing to control, Example: a) severe infection occurred within 4 weeks before initiation of study treatment, Including but not limited to hospitalization for infection, bacteremia or complications of severe pneumonia; Or having received therapeutic oral or intravenous antibiotics within two weeks prior to starting study treatment, Patients receiving prophylactic antibiotic therapy may be enrolled (e. g. prevention of urinary tract infection or chronic obstructive pulmonary disease); b) symptomatic congestive heart failure (New York Heart Association Grade II-IV) or symptomatic or poorly controlled arrhythmia; c) with other malignancies within 5 years prior to treatment (cutaneous carcinoma, breast / cervix, and in situ, nonmelanoma with radical treatment and no evidence of disease recurrence); And d) suspected or confirmed subjects with acute promyelocytic leukemia (indicated by morphology, immunotyping, molecular testing, or chromosome karyotype); e) subjects with current cancerous meningitis, spinal cord compression, etc.; f) a history of poorly controlled hypertension and diabetes; g) symptomatic endogenous lung disease; h) any arterial thromboembolic event within 6 months prior to inclusion, Including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack; i) significant malnutrition, If intravenous nutrition solution is needed. Stable for more than 4 weeks after correction of malnutrition before the first dose of study drug can be enrolled; j) tumor invasion of important surrounding organs or blood vessels (such as mediastinal macrovessels, superior vena cava, trachea, esophagus, etc.), Or at risk of oesophageal tracheal fistula or oesophageal pleural fistula; k) after esophageal or endotracheal cavity stenting; l) other acute or chronic diseases or abnormal laboratory test values that may lead to the following results: increase the risk associated with study participation or study drug administration, Or to interfere with the interpretation of the study findings, And listed the subject as ineligible for the study at the discretion of the investigator; m) a history of gastrointestinal perforation and / or fistula within 6 months prior to study inclusion. N) with an uncontrolled third-space effusion requiring repeated drainage, such as pleural fluid, ascites, and pericardial effusion.(Patients who do not require drainage or have no significant increase for 3 days can be enrolled).

   9. Patients with active gastrointestinal or other diseases, as well as factors such as surgical resection that may significantly affect drug absorption, metabolism, or excretion. Including but not limited to the following situations: malabsorption syndrome, inflammatory bowel disease, partial or complete intestinal obstruction, gastric or small intestine resection surgery.

   10. Patients had a history of severe underlying pulmonary disease or medical conditions, such as moderate to severe chronic obstructive pulmonary disease (COPD), interstitial pulmonary disease (ILD), drug-induced ILD, acute or chronic infectious pneumonia, lung transplantation, etc.; 11. Pregnant or lactating women. 12 is participating in another interventional clinical study and has not completed study treatment.

   13 A known history of allogeneic organ transplantation and allogeneic HSCT. 14. Major surgical procedure (craniotomy, thoracotomy, laparotomy, vascular intervention, otherwise defined by the investigator) within 4 weeks of the first administration of the study drug, or the presence of an unhealed wound, ulcer, or fracture. Note: Local surgical treatment of isolated lesions is acceptable for the purpose of palliative treatment.

   15. HIV-infected persons (HIV 1 / 2 antibody-positive). 16 Known active syphilis infection, active pulmonary tuberculosis. 17 Patients with a clear history of mental disorders and medication for treatment.

   18. People with a history of drug abuse or drug use. 19. The investigator considers that the patient has other factors that may affect the study results and interfere with the entire study process, including previous, or existing physical conditions, treatment or laboratory abnormalities, and the subject's unwillingness to comply with the procedures, limitations and requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | each cycle is 21 or28 days,from the first use until the date of first documented progression or date of death from any cause or start new anti-tumor therapy or withdraw ICF or the study is over，whichever came first, assessed up to 24 months
  ORR based on molecular subtyping of small cell lung cancer

IPD SHARING:
Plan to Share IPD: No